CLINICAL TRIAL: NCT05601765
Title: The Effect of Digital Team-based Communication Between Orthopaedic Surgery Patients and Healthcare Professionals on Patient-initiated Telephone Contacts to Hospital After Discharge: a Randomized Controlled Trial
Brief Title: The Effect of Digital Team-based Communication on Patient-initiated Telephone Contacts to Hospital After Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Ole Rahbek, Professor, MD, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-219
Record Dates: First submitted 2022-10-28; First posted 2022-11-01 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Orthopaedic Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard communication pathways after discharge (Active Comparator): Patients who need contact within 72 hours of discharge are advised to call the bed section, from where they were discharged. Telephone counseling can be provided by the nurses available at the time of calling (e.g., questions for medical treatment, precautions after surgery etc.).
  * If deemed relevant, the patient may be asked to appear in person at the ward (e.g., for the examination of wounds).
  * If more serious conditions are suspected, a doctor or emergency department will be contacted by the nurse for assessment, triage and possibly readmission.
  Patients who need contact after 72 hours of discharge are advised to call the outpatient clinic, if they have planned attendances here, or alternatively their own general practitioner or home care nurse.
  Standard communication pathways between healthcare professionals across sectors are electronic correspondences and telephone inquiries.
  Interventions: Other: Standard communication pathways after discharge
- Digital team-based communication after discharge (Experimental): Patients will be given access to digital communication with their healthcare team across sectors who are involved in their treatment and care after hospital discharge (eDialogue). They will be set up in a messenger-like tool on the day of discharge, and relevant healthcare professionals will be connected. Individually, the patients will define who they would like to involve, and consent is given digitally. The minimum participants for each patient will be the patient and/or their closest relative, the orthopaedic surgeon, a nurse from the outpatient clinic and a secretary. Patients will have access to eDialogue for 60 days after discharge, and the response rate is set to be 24 hours on weekdays. On weekends and public holidays, patients are informed that they cannot expect a response. If the primary healthcare professional is registered to be on vacation or other absence, "substitutes" within the respective health professional groups will be included.
  Interventions: Other: Digital team-based communication after discharge

INTERVENTIONS:
Other: Standard communication pathways after discharge — Standard communication pathways after discharge
  Arms: Standard communication pathways after discharge
Other: Digital team-based communication after discharge — Standard communication pathways plus digital team-based communication after discharge
  Arms: Digital team-based communication after discharge

SUMMARY:
The aim of this study is to investigate the effects of eDialogue versus standard communication pathways on patient-initiated telephone contacts to the hospital following discharge. Secondary aims are to explore the effect on other patient-initiated contacts after hospital discharge (mail, video, SMS, personal attendance) and, if digital team-based communication can positively affect patients experience of continuity of care.

DETAILED DESCRIPTION:
Transition of care from hospital to home following orthopaedic surgery pose a significant risk to patient safety. After discharge, patients or primary care providers may need to communicate with the specialized healthcare team at the hospital about symptoms, postoperative complications, rehabilitation, wounds and medication, but are hampered by a fragmented healthcare system with slow communication pathways. Communication through phone often involves several intermediaries and waiting time for both patients and healthcare professionals. The fact that patients and healthcare professionals must be present at the same time is inflexible and disruptive to work processes. However, cross-sectoral communication and collaboration with patients after hospital discharge are prerequisites to achieve high-quality care and good patient outcomes. Review of the literature show that few studies have explored the effects of digital team-based communication with the patient and across sectors to facilitate collaboration and knowledge sharing after discharge. On the basis of findings from a preliminary pilot study suggesting asynchronous digital team-based communication between orthopaedic surgery patients and healthcare professionals across sectors (eDialogue) may be a solution to the existing problems in communication pathways, we initiated this trial.

ELIGIBILITY:
Patients are recruited from the following orthopaedic surgery sub-specialties at Aalborg University Hospital:

* Deformity surgery
* Trauma surgery, including fractures of the spine

Inclusion Criteria:

Patients admitted and operated at Aalborg University Hospital, who;

* have complex care needs involving cross disciplinary and cross sectoral care after hospital discharge
* will be discharged to their home
* will need follow-up in the outpatient clinic after discharge

Patients at all ages, but:

* if patient is < 15 years old, the parent(s) will be included in the study as user(s) of LetDialog.
* if patient is 15-18 years old, the patient will be the user in LetDialog and answer the questionnaires to comply with existing Danish legislation Health Act § 17. If the patient wishes, parent(s) can be included as user(s) in LetDialog as well.

Have access to and ability to use a smartphone Have access to NemID (needed to create a GDPR-safe user profile in LetDialog)

Exclusion Criteria:

Patients, who:

* have previously participated in the eDialogue pilot study
* are discharged to a rehabilitation center, nursing home or similar
* do not speak/read Danish or English well enough to understand participant information and use digital communication in Danish or English through LetDialog
* are included in other ongoing randomized controlled trials or prospective follow-up studies in the Orthopaedic Surgery Department at Aalborg University Hospital, where participation could possibly affect the results of these studies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Patient-initiated telephone contacts to hospital up to 8 weeks after discharge | 8 weeks
  Questionnaire on patient-initiated telephone contacts to hospital after discharge distributed once a week for 8 weeks after discharge. The questionnaire is short, self-developed and not validated, but tested for wording and understanding in 12 orthopaedic surgery patients using qualitative interviewing.

SECONDARY OUTCOMES:
Other patient-initiated contacts to hospital or other healthcare facilities through email, video, SMS up to 8 weeks after discharge | 8 weeks
  Questionnaire on patient-initiated contacts to hospital or other healthcare facilities after discharge through email, video, SMS distributed on once a week for 8 weeks after discharge. The questionnaire is self-developed and not validated, but tested for wording and understanding in 12 orthopaedic surgery patients using qualitative interviewing.
Patient Continuity of Care | 4 weeks
  Validated questionnaire containing 41 items. 27 items belong to 'before discharge' and will be administered on the day of discharge and 14 items belong to 'after discharge' and will be administered 30 days after discharge.
Feeling safe and satisfied with access to healthcare professionals | 8 weeks
  Questionnaire to test if intervention provides feeling of safety and satisfaction with access to healthcare professionals after discharge. The questionnaire is self-developed to fit the intervention. It contains of 4 items for the control group and 7 items for the intervention group and will be distributed 8 weeks after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Ole Rahbek, PhD, MD, Principal Investigator — Interdisciplinary Orthopaedics, Aalborg University Hospital, Denmark; Lili WH Jensen, MSc, Study Chair — Interdisciplinary Orthopaedics, Aalborg University Hospital, Denmark; Birthe I Dinesen, PhD, MSc, Study Chair — Aalborg University; Søren Kold, PhD, MD, Study Chair — Interdisciplinary Orthopaedics, Aalborg University Hospital, Denmark
Locations (1):
- Orthopaedic Surgery Department, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After 1 year from study start
Access Criteria: Researchers that provide a methodologically sound plan